CLINICAL TRIAL: NCT03084770
Title: A Prospective Evaluation of the Management of Sporadic Asymptomatic Nonfunctioning Pancreatic Neuroendocrine Neoplasms ≤ 2 cm
Brief Title: Asymptomatic Small Pancreatic Endocrine Neoplasms.
Acronym: ASPEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Falconi, full Professor, IRCCS San Raffaele
Other Study IDs: ASPEN
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Non Functioning Pancreatic Endocrine Tumor
Keywords: NF-PNEN
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active surveillance group: Advised surveillance strategy consists of imaging studies (MR or EUS or US), every 6 months for the first two years and yearly thereafter for five years in the absence of significant changes on imaging or symptoms appearance. During surveillance, a high-quality imaging technique (MRI or CT) is mandatory at least every 12 months. Determination of CgA during follow-up is at physician's discretion. During follow-up, the treating physician is responsible for patient management and decision-making.
  Interventions: Diagnostic Test: Radiological imaging studies; Other: Quality of Life Assessment
- Surgical resection group: Timing and type of resection will be established by the treating physician. Follow up strategy after surgery consists of imaging studies (MR or CT), every 6 months for the first two years and yearly thereafter for five years. An high-quality imaging technique (MRI or CT) is mandatory at least every 12 months. Determination of CgA during follow-up is at physician's discretion. During follow-up, the treating physician is responsible for patient management and decision-making. Date of surgery does not change the timing of follow up which starts from the date of enrolment.
  Interventions: Diagnostic Test: Radiological imaging studies; Other: Quality of Life Assessment

INTERVENTIONS:
Diagnostic Test: Radiological imaging studies — Patients will be submitted to radiological imaging studies (CT scan and/or MRI and/ or 68Gallium PET/CT and/or Octreoscan and/or EUS+FNAand/or Octreoscan and/or EUS+FNA) at diagnosis, and then every 6 months for the first two years and yearly thereafter for five years in the absence of significant changes on imaging or symptoms appearance. Every 12 months (or 6 months for patients with Ki67> 2%) a high quality imaging (CT scan or MRI) is required.
Other: Quality of Life Assessment — quality of life and the perceived burden of surveillance or follow-up after surgery for participants, will be investigated by administrating HADS questionnaire and EORTC QLQ-C30 (version 3) and EORTC QLQ-GI.NET21 Module.

SUMMARY:
The aim of the study is to evaluate the most appropriate management of sporadic asymptomatic non-functioning pancreatic neuroendocrine neoplasms (NF-PNEN) ≤ 2 cm. P NF-PNEN management will be decided at the hospital and all therapeutics decision will be decided/coordinated by the treating physician.

Patients will be either submitted to surgical resection or to active surveillance.

DETAILED DESCRIPTION:
In the last decade a dramatic increase in diagnosis of small, incidentally discovered, NF-PNEN was observed. Various study indicates the safety of a conservative management for this lesion and the The European Neuroendocrine Tumor Society (ENETS) proposed a "wait and see" approach for small NF-PNEN.

Indications for surgery include the presence of a localized NF-PNEN in the absence of distant metastases as curative resection of these tumors is associated with favourable prognosis especially for low grade.

In the last decade a dramatic increase in diagnosis of small, incidentally discovered, NF-PNEN was observed.Moreover, other investigators observed a clear relationship between the tumor diameter and low risk of malignancy and systemic progression.

In particular, a tumor size ≤ 2 cm seems to be associated with a negligible risk of disease recurrence and with a very low incidence of aggressive features such as lymph node involvement.On this basis, the European Neuroendocrine Tumor Society (ENETS) proposed a "wait and see" approach for small NF-PNEN when incidentally discovered. Since then, various series evaluated the safety of a conservative management for small, sporadic, incidentally diagnosed, NF-PNEN.

After a median follow-up of 28-45 months, all the studies confirmed that an intensive surveillance for incidental and small NF-PNEN is safe in selected cases.

Nevertheless, available data are based only on retrospective series with a significant heterogeneity of inclusion criteria and different tumor diameter cut-off and the appropriate management of this entities (surveillance versus surgery) is still a matter of debate.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Individuals with asymptomatic sporadic NF-PNEN ≤ 2 cm
* Diagnosis has to be proven by a positive fine-needle aspiration (FNA) or by the presence of a measurable nodule on high-quality imaging technique (CT or MR) that is positive at 68Gallium DOTATOC-PET scan or Octreoscan.
* Patients who undergo surgery for NF-PNEN<2cm within 12 months. In these cases, diagnosis has to be proven by histological confirmation of NF-PNEN
* Informed consent

Exclusion Criteria:

* NF-PNEN > 2 cm of maximum diameter
* Presence of genetic syndrome (MEN1, VHL, NF)
* Presence of symptoms (specific symptoms suspicious of a clinical syndrome related to hypersecretion of bioactive compounds) or unspecific symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a newly diagnosis (less thn 12 months) of non- functioning pancreatic endocrine neoplasia (NF-PNEN) ≤ 2 cm of diameter. Either patients submitted to surgery or in active surveillance can be enrolled. Patients with sindrome or genetics disorders are excluded from the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease/progression-free survival of NF-PNEN ≤ 2 cm | From date of enrolment until the date of first documented progression or first evidence of recurrence, from 6 months up to 6 years.
  The primary endpoint is disease/progression-free survival, defined as the time from study enrolment to the first evidence of progression (active surveillance group) or recurrence of disease (surgical resection group) or death from disease.

SECONDARY OUTCOMES:
Frequency of NF-PNEN ≤ 2 cm | 6 years
  The secondary end point is to evaluate the frequency of asymptomatic sporadic NF-PNEN ≤ 2 cm among overall sporadic NF-PNEN. Participating centers are required to give yearly the number of patients with NF-PNEN referred to their institution.
Outcome of surgical intervention of NF-PNEN ≤ 2 cm | from the date of surgery to 1 months later the surgery
  Morbidity and mortality of patients submitted to surgical resection
Epidemiology of patients submitted to surgical intervention for NF-PNEN ≤ 2 cm | from the date of surgery, up to 6 years
  Number of patients submitted to surgery andh type of surgical procedures.
Evolution of NF-PNEN ≤ 2 cm | From date of enrolment until the date of first documented radiological evolution, from 6 months up to 6 years.
  NF-PNEN evolution, in terms of development of symptoms, tumour growth, development of distant metastases and secondary pancreatic duct dilatation.
Quality of Life of NF-PNEN ≤ 2 cm | from 6 months up to 6 years.
  The perceived burden of surveillance or follow-up after surgery for participants, as assessed by questionnaires regarding attitude towards surveillance and general anxiety and depression (Hospital Anxiety and Depression scale, HADS). Quality of Life will be investigated, by filling in EORTC QLQ-C30 (version 3) and EORTC QLQ-GI.NET21 Module.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Falconi, Professor, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falconi M, Eriksson B, Kaltsas G, Bartsch DK, Capdevila J, Caplin M, Kos-Kudla B, Kwekkeboom D, Rindi G, Kloppel G, Reed N, Kianmanesh R, Jensen RT; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for the Management of Patients with Functional Pancreatic Neuroendocrine Tumors and Non-Functional Pancreatic Neuroendocrine Tumors. Neuroendocrinology. 2016;103(2):153-71. doi: 10.1159/000443171. Epub 2016 Jan 5. No abstract available. PMID 26742109
- [Background] Jilesen AP, van Eijck CH, Busch OR, van Gulik TM, Gouma DJ, van Dijkum EJ. Postoperative Outcomes of Enucleation and Standard Resections in Patients with a Pancreatic Neuroendocrine Tumor. World J Surg. 2016 Mar;40(3):715-28. doi: 10.1007/s00268-015-3341-9. PMID 26608956
- [Background] Hashim YM, Trinkaus KM, Linehan DC, Strasberg SS, Fields RC, Cao D, Hawkins WG. Regional lymphadenectomy is indicated in the surgical treatment of pancreatic neuroendocrine tumors (PNETs). Ann Surg. 2014 Feb;259(2):197-203. doi: 10.1097/SLA.0000000000000348. PMID 24253141
- [Background] Kuo EJ, Salem RR. Population-level analysis of pancreatic neuroendocrine tumors 2 cm or less in size. Ann Surg Oncol. 2013 Sep;20(9):2815-21. doi: 10.1245/s10434-013-3005-7. Epub 2013 Jun 15. PMID 23771245
- [Background] Vagefi PA, Razo O, Deshpande V, McGrath DJ, Lauwers GY, Thayer SP, Warshaw AL, Fernandez-Del Castillo C. Evolving patterns in the detection and outcomes of pancreatic neuroendocrine neoplasms: the Massachusetts General Hospital experience from 1977 to 2005. Arch Surg. 2007 Apr;142(4):347-54. doi: 10.1001/archsurg.142.4.347. PMID 17438169
- [Background] Crippa S, Partelli S, Zamboni G, Scarpa A, Tamburrino D, Bassi C, Pederzoli P, Falconi M. Incidental diagnosis as prognostic factor in different tumor stages of nonfunctioning pancreatic endocrine tumors. Surgery. 2014 Jan;155(1):145-53. doi: 10.1016/j.surg.2013.08.002. PMID 24646958
- [Background] Birnbaum DJ, Gaujoux S, Cherif R, Dokmak S, Fuks D, Couvelard A, Vullierme MP, Ronot M, Ruszniewski P, Belghiti J, Sauvanet A. Sporadic nonfunctioning pancreatic neuroendocrine tumors: prognostic significance of incidental diagnosis. Surgery. 2014 Jan;155(1):13-21. doi: 10.1016/j.surg.2013.08.007. Epub 2013 Nov 12. PMID 24238123
- [Background] Bettini R, Partelli S, Boninsegna L, Capelli P, Crippa S, Pederzoli P, Scarpa A, Falconi M. Tumor size correlates with malignancy in nonfunctioning pancreatic endocrine tumor. Surgery. 2011 Jul;150(1):75-82. doi: 10.1016/j.surg.2011.02.022. PMID 21683859
- [Background] Haynes AB, Deshpande V, Ingkakul T, Vagefi PA, Szymonifka J, Thayer SP, Ferrone CR, Wargo JA, Warshaw AL, Fernandez-del Castillo C. Implications of incidentally discovered, nonfunctioning pancreatic endocrine tumors: short-term and long-term patient outcomes. Arch Surg. 2011 May;146(5):534-8. doi: 10.1001/archsurg.2011.102. PMID 21576607
- [Background] Cherenfant J, Stocker SJ, Gage MK, Du H, Thurow TA, Odeleye M, Schimpke SW, Kaul KL, Hall CR, Lamzabi I, Gattuso P, Winchester DJ, Marsh RW, Roggin KK, Bentrem DJ, Baker MS, Prinz RA, Talamonti MS. Predicting aggressive behavior in nonfunctioning pancreatic neuroendocrine tumors. Surgery. 2013 Oct;154(4):785-91; discussion 791-3. doi: 10.1016/j.surg.2013.07.004. PMID 24074416
- [Background] Partelli S, Gaujoux S, Boninsegna L, Cherif R, Crippa S, Couvelard A, Scarpa A, Ruszniewski P, Sauvanet A, Falconi M. Pattern and clinical predictors of lymph node involvement in nonfunctioning pancreatic neuroendocrine tumors (NF-PanNETs). JAMA Surg. 2013 Oct;148(10):932-9. doi: 10.1001/jamasurg.2013.3376. PMID 23986355
- [Background] Falconi M, Bartsch DK, Eriksson B, Kloppel G, Lopes JM, O'Connor JM, Salazar R, Taal BG, Vullierme MP, O'Toole D; Barcelona Consensus Conference participants. ENETS Consensus Guidelines for the management of patients with digestive neuroendocrine neoplasms of the digestive system: well-differentiated pancreatic non-functioning tumors. Neuroendocrinology. 2012;95(2):120-34. doi: 10.1159/000335587. Epub 2012 Feb 15. No abstract available. PMID 22261872
- [Background] Gaujoux S, Partelli S, Maire F, D'Onofrio M, Larroque B, Tamburrino D, Sauvanet A, Falconi M, Ruszniewski P. Observational study of natural history of small sporadic nonfunctioning pancreatic neuroendocrine tumors. J Clin Endocrinol Metab. 2013 Dec;98(12):4784-9. doi: 10.1210/jc.2013-2604. Epub 2013 Sep 20. PMID 24057286
- [Background] Lee LC, Grant CS, Salomao DR, Fletcher JG, Takahashi N, Fidler JL, Levy MJ, Huebner M. Small, nonfunctioning, asymptomatic pancreatic neuroendocrine tumors (PNETs): role for nonoperative management. Surgery. 2012 Dec;152(6):965-74. doi: 10.1016/j.surg.2012.08.038. Epub 2012 Oct 24. PMID 23102679
- [Background] Jung JG, Lee KT, Woo YS, Lee JK, Lee KH, Jang KT, Rhee JC. Behavior of Small, Asymptomatic, Nonfunctioning Pancreatic Neuroendocrine Tumors (NF-PNETs). Medicine (Baltimore). 2015 Jul;94(26):e983. doi: 10.1097/MD.0000000000000983. PMID 26131843
- [Background] Sadot E, Reidy-Lagunes DL, Tang LH, Do RK, Gonen M, D'Angelica MI, DeMatteo RP, Kingham TP, Groot Koerkamp B, Untch BR, Brennan MF, Jarnagin WR, Allen PJ. Observation versus Resection for Small Asymptomatic Pancreatic Neuroendocrine Tumors: A Matched Case-Control Study. Ann Surg Oncol. 2016 Apr;23(4):1361-70. doi: 10.1245/s10434-015-4986-1. Epub 2015 Nov 23. PMID 26597365
- [Background] Rosenberg AM, Friedmann P, Del Rivero J, Libutti SK, Laird AM. Resection versus expectant management of small incidentally discovered nonfunctional pancreatic neuroendocrine tumors. Surgery. 2016 Jan;159(1):302-9. doi: 10.1016/j.surg.2015.10.013. Epub 2015 Nov 4. PMID 26547726
- [Background] Partelli S, Cirocchi R, Crippa S, Cardinali L, Fendrich V, Bartsch DK, Falconi M. Systematic review of active surveillance versus surgical management of asymptomatic small non-functioning pancreatic neuroendocrine neoplasms. Br J Surg. 2017 Jan;104(1):34-41. doi: 10.1002/bjs.10312. Epub 2016 Oct 5. PMID 27706803
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Yadegarfar G, Friend L, Jones L, Plum LM, Ardill J, Taal B, Larsson G, Jeziorski K, Kwekkeboom D, Ramage JK; EORTC Quality of Life Group. Validation of the EORTC QLQ-GINET21 questionnaire for assessing quality of life of patients with gastrointestinal neuroendocrine tumours. Br J Cancer. 2013 Feb 5;108(2):301-10. doi: 10.1038/bjc.2012.560. Epub 2013 Jan 15. PMID 23322194
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Derived] Partelli S, Ramage JK, Massironi S, Zerbi A, Kim HB, Niccoli P, Panzuto F, Landoni L, Tomazic A, Ibrahim T, Kaltsas G, Bertani E, Sauvanet A, Segelov E, Caplin M, Coppa J, Armstrong T, Weickert MO, Butturini G, Staettner S, Boesch F, Cives M, Moulton CA, He J, Selberherr A, Twito O, Castaldi A, De Angelis CG, Gaujoux S, Almeamar H, Frilling A, Vigia E, Wilson C, Muffatti F, Srirajaskanthan R, Invernizzi P, Lania A, Kwon W, Ewald J, Rinzivillo M, Nessi C, Smid LM, Gardini A, Tsoli M, Picardi EE, Hentic O, Croagh D, Toumpanakis C, Citterio D, Ramsey E, Mosterman B, Regi P, Gasteiger S, Rossi RE, Smiroldo V, Jang JY, Falconi M. Management of Asymptomatic Sporadic Nonfunctioning Pancreatic Neuroendocrine Neoplasms (ASPEN) </=2 cm: Study Protocol for a Prospective Observational Study. Front Med (Lausanne). 2020 Dec 23;7:598438. doi: 10.3389/fmed.2020.598438. eCollection 2020. PMID 33425946